CLINICAL TRIAL: NCT00318201
Title: The Effect of Concomitant Administration of Erythromycin and Diltiazem on CYP3A Activity in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Stephen D. Hall, Indiana University
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: # 0412-09; R01GM067308/NIGMS; MO1RR000750/GCRC #1267; R01GM067308 (NIH)
Record Dates: First submitted 2006-04-21; First posted 2006-04-26 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Erythromycin; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Altered efficacy for drug to drug interaction of diltiazam with erythromycin
  Interventions: Drug: Erythromycin; Drug: Diltiazem

INTERVENTIONS:
Drug: Erythromycin
Drug: Diltiazem

SUMMARY:
We, the researchers at the Indiana University School of Medicine, are doing this study to better understand how the effects of certain medications are altered when taken simultaneously, or in combination with each other. We will also look at how each volunteer's genes (DNA) may affect the way these medications are metabolized.

Hypothesis:

We will test the hypothesis that the extent of drug-drug interaction caused by the combination of erythromycin and diltiazem is not predictable from the extent of interaction produced by each inhibitor alone. Specifically we will test the hypothesis that the combination of erythromycin and diltiazem will cause a greater decrease in midazolam intravenous and oral clearance than the sum of the decreases caused by each inhibitor alone.

DETAILED DESCRIPTION:
Many drugs such as diltiazem are metabolized by CYP3A4, the cytochrome P450 enzyme responsible for the metabolism of erythromycin and when given together, the possibility exists that one drug inhibits the metabolism of the other leading to an increase in plasma concentration. The magnitude of this interaction is not known. It is therefore important to define this effect because diltiazem is a drug that is used commonly to treat hypertension, angina and atrial fibrillation and these patients may be given erythromycin for the treatment of intercurrent bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

Approximately 45 healthy volunteers may be recruited to participate in the study, with a goal of 15 healthy volunteers (7 or 8 males) completing the entire four phases. All potential subjects:

1. Must be a non-smoker
2. Between 18 to 50 years of age
3. Have a body mass index of 30 or less
4. Must be willing to undergo a screening physical examination and proven to be free from metabolic, cardiac, pulmonary, renal or hepatic dysfunction as determined by the screening physical, medical history, 12-lead electrocardiography, and laboratory values which include: a CMP (complete metabolic profile), a CBC/diff/plt (complete blood count with differential and platelet count), serum pregnancy test (if applicable), and UA (urinalysis). Also, given the uncertain effects of these drugs on the fetus and the fact that hormonal contraceptives are prohibited, the female subjects should be on two other forms of birth control (e.g. condom, contraceptive foam).

Exclusion Criteria:

Potential volunteers will be excluded:

1. If they have allergies or are hypersensitive to any of the study medications:

   A. Midazolam (Versed) or related benzodiazepines drugs such as diazepam (Valium) or alprazolam (Xanax).

   B. Diltiazem (Cardizem, Dilacor) or related calcium channel blockers such as verapamil (Calan, Isoptin).

   C. Erythromycin (Erythrocin, E-mycin, Ery-tab) or related antibiotics such as clarithromycin (Biaxin) or have experienced abdominal pain when taking erythromycin or other related medications.
2. If they are taking any prescription medication on a regular basis including contraceptives such as oral birth control pills, transdermal patches or injections (Depo-Provera).
3. If they are taking over-the-counter medications, any herbal or dietary supplement (including Benadryl, Sudafed, St. John's wort, herbal teas, vitamins and garlic supplements) that cannot be stopped for the study duration. Use of over-the-counter drugs for the treatment of minor, short-lived (2 to 3 days) symptoms may be allowable (such as Tylenol) but must first be approved by a study investigator.
4. If they have donated blood within the past two months, or are anemic (have a hemoglobin level less than 12.5 mg/dl).
5. If they weigh less than 52 kg, or have a BMI (Body Mass Index) greater than 32.
6. If they have a screening or baseline EKG reading that is abnormal or could place them at higher risk as decided by the study doctors (baseline corrected QT interval in the EKG of 450 msec or greater or a baseline PR interval in the EKG of 210 msec or greater).
7. If they have a history of bradycardia or consistently have a heart rate less than 55 beats per minutes.
8. If they have any history of heart disease or have a family medical history of sudden death (heart stopping suddenly without warning).
9. If they have a history of psychiatric problems that may be exacerbated by participation in this study, or if the subject can not state a good understanding of this study's risks and requirements.
10. If they have a positive serum pregnancy test during the screening process or have a positive urine pregnancy test (UPT) which will be obtained just prior to each of the four study phases.
11. If they are currently breastfeeding.
12. If they have participated in any other study in which they have taken a research medication within the past three months.
13. If they have a history of alcohol or drug abuse, or have used tobacco or marijuana within the past three months.
14. If they are unwilling or unable to refrain from using drugs, alcohol, or any food listed on the exclusion list below during this study.
15. If they are an employee or student under the supervision of any study investigator.
16. If they are unwilling or unable to follow the study rules.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2006-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Primary Aims: To quantify the extent of the drug-drug interaction between erythromycin and midazolam | 2 days
To quantify the extent of the drug-drug interaction between diltiazem and midazolam | 2 days
To quantify the extent of the drug-drug interaction between the combination of diltiazem and erythromycin, and midazolam | 2 days

SECONDARY OUTCOMES:
Secondary Aims: To quantify the effects of erythromycin, diltiazem, and the combination of erythromycin and diltiazem on the electrocardiogram (EKG) PR interval | 2 days
To quantify the effects of erythromycin, diltiazem, and the combination of erythromycin and diltiazem on the heart-rate corrected QT interval of the EKG | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Hall, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Medical Center / GCRC, Indianapolis, Indiana, United States